CLINICAL TRIAL: NCT06710379
Title: A Phase 1a/b Study of ADRX-0405 in Subjects With Select Advanced Solid Tumors
Brief Title: A Study of ADRX-0405 in Subjects With Select Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Adcentrx Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADRX-0405-001
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-11

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1a Dose Escalation (Experimental): Increasing doses of ADRX-0405 will be administered to identify the maximum tolerated dose (MTD) and the recommended dose to be used in the Phase 1b part.
  Interventions: Drug: ADRX-0405
- Phase 1b Dose Expansion (Experimental): ADRX-0405 will be initially administered at the dose recommended from the Phase 1a part in subjects with previously treated mCRPC.
  Interventions: Drug: ADRX-0405

INTERVENTIONS:
Drug: ADRX-0405 — Antibody Drug Conjugate targeting STEAP1

SUMMARY:
The primary purpose of this study is to assess the safety, tolerability, and pharmacokinetics, and to identify the optimal dose of ADRX-0405 in patients with select advanced solid tumors.

DETAILED DESCRIPTION:
This is a 2-part study. The Phase 1a will consist of a dose escalation of ADRX-0405 to evaluate initial safety and tolerability in patients with select advanced solid tumors [including metastatic castration resistant prostate cancer (mCRPC), gastric cancer (GC), and non-small cell lung cancer (NSCLC)], and to identify the recommended dose to be used in the Phase 1b. The Phase 1b will further evaluate the safety and tolerability, as well as preliminary efficacy, and identify the optimal dose of ADRX-0405 in subjects with previously treated metastatic castration resistant prostate cancer (mCRPC).

ELIGIBILITY:
Inclusion Criteria:

* Phase 1a Dose Escalation: Subjects with histologically confirmed select advanced solid tumors, including metastatic castration resistant prostate cancer (mCRPC), gastric cancer (GC), and non-small cell lung cancer (NSCLC).
* Phase 1b Dose Expansion: Subjects with histologically confirmed prostate adenocarcinoma that is confirmed to be castration resistant (i.e., serum testosterone < 50 ng/dL [< 2.0 nM]) and that is intolerant/resistant to standard of care (SOC) therapies.
* Measurable disease according to RECIST version 1.1 or evaluable disease per PCWG3 for subjects with prostate cancer
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 in 1a; 0-2 in 1b
* Adequate hematologic, liver, and renal function

Exclusion Criteria:

* Active and uncontrolled central nervous system metastases
* Significant cardiovascular disease
* History of another malignancy other than the one for which the subject is being treated on this study within 3 years
* Receipt of any anticancer or investigational therapy within: 5 elimination half-lives or 14 days (whichever is less); 4 weeks for any therapeutic radiopharmaceutical for prostate cancer
* History of (non-infectious) ILD/pneumonitis that required steroids within 2 years of study enrollment, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Receiving systemic antimicrobial treatment for active infection; routine antimicrobial prophylaxis is permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Until study completion (estimated 2 years)

SECONDARY OUTCOMES:
Measurement of End of Infusion or observed maximum blood concentration (Ceoi orCmax) of ADRX-0405 | Until study completion (estimated 2 years)
  Measured from pharmacokinetic (PK) blood samples
Measurement of trough concentration (Ctrough) of ADRX-0405 | Until study completion (estimated 2 years)
  Measured from PK blood samples
Measurement of area under the blood concentration-time curve (AUC) of ADRX-0405 | Until study completion (estimated 2 years)
  Measured from PK blood samples
Measurement of partial area under the concentration-time curve after first dose (AUC0-21) of ADRX-0405 and as appropriate | Until study completion (estimated 2 years)
  Measured from PK blood samples
Measurement of terminal or apparent terminal half-life (t1/2) of ADRX-0405 | Until study completion (estimated 2 years)
  Measured from PK blood samples
Measurement of systemic clearance (CL) and volume of distribution at steady state (Vss) as appropriate of ADRX-0405 | Until study completion (estimated 2 years)
  Measured from PK blood samples
Incidence of anti-drug antibody (ADA) to ADRX-0405 | Until study completion (estimated 2 years)
  Measured from ADA blood samples
Measurement of objective response rate (ORR) per RECIST 1.1 | Until study completion (estimated 2 years)
  Percentage of subjects achieving complete response (CR) or partial response (PR)
ORR per Prostate Cancer Working Group 3 (PCWG3) | Until study completion (estimated 2 years)
  Percentage of subjects achieving complete response (CR) or partial response (PR)
Measurement of duration of response (DOR) | Until study completion (estimated 2 years)
  Time from first response until first evidence of disease progression (PD) or death from any cause
Measurement of disease control rate (DCR) | Until study completion (estimated 2 years)
  Percentage of subjects achieving CR, PR or stable disease (SD)
Measurement of progression free survival (PFS) | Until study completion (estimated 2 years)
  Time from the start of study drug until first evidence of PD or death from any cause
Measurement of radiographic progression free survival (rPFS) | Until study completion (estimated 2 years)
  Time from the start of study drug until first radiographic documentation of PD, or death from any cause, whichever comes first
Measurement of overall survival (OS) | Until study completion (estimated 2 years)
  Time from the start of study drug until death from any cause

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - City of Hope, Duarte, California
  - UCLA, Santa Monica, California
  - START Midwest, Grand Rapids, Michigan
  - University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - NEXT Austin, Austin, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - START Mountain Region, West Valley City, Utah
  - NEXT Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No